CLINICAL TRIAL: NCT05495867
Title: Evaluation of a Bioactive Surface in Post-extraction Sites: Case Control Study
Brief Title: Evaluation of Implant-prosthetic Rehabilitation Performed With Two Implants With Different Surface Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luigi Canullo (Other)
Responsible Party: Sponsor-Investigator, Luigi Canullo, Principal investigator, Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo
Organization: Studio Odontoiatrico Associato Dr. P. Cicchese e L. Canullo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABT1
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Missing Teeth; Edentulous Jaw; Edentulous Mouth
Keywords: dental implant; bioactivation; implant surface
MeSH Terms: conditions — Anodontia; Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NINA- MultiNeO NH (Experimental): implant with bioactive surface
  Interventions: Procedure: implant placement
- MultiNeO CS (Active Comparator): implant with traditional surface
  Interventions: Procedure: implant placement

INTERVENTIONS:
Procedure: implant placement — implant placement in edentulous area

SUMMARY:
In this case-control study a bioactive implant surface was compared with traditional surfaced implants. Primary objectives: Test the implant stability in post-extractive sites, comparing traditional surfaced implants (MultiNeO CS, control group) to bioactive surfaced implants (NINA- MultiNeO NH, treatment group).

Primary outcome endpoints were Implant stability, assessed through Implant stability quotient (ISQ) values and Marginal bone loss (MBL)

DETAILED DESCRIPTION:
In this post- market case control study, the tested CE-marked dental implants are MultiNeO CS 1930 and NINA MultiNeO NH 9330, both manufactured by Alpha-Bio Tec. .

Alpha-Bio Tec. implants systems are made of Ti-6AI-4V ELI Titanium alloy which is a high-performance and highly biocompatible alloy for manufacturing bone implants. Alpha-Bio Tec developed the superior NanoTec&trade implant surface for optimized osseointegration process. Alpha-Bio Tec NanoTec™ implant surface is achieved by a complex process of large particle sandblasting and acid etching. Sandblasting with large particles allows the creation of macropores (20-40 microns), while the double etching allows the creation of micropores (1-5 microns). The micro - structure and roughness properties of NanoTec™ Implant Surface greatly influences the dynamic wettability of implant surfaces during the initial contact with the host.

The overwritten implant surface enables greater absorption of blood and plasma proteins directly inside the micropores, immediately after the implant has been placed.

It is the implant surface of MultiNeO. NeO or MultiNeO is defined as a system since it includes three types of connections: a conical narrow connection (CHC), a conical standard conical connection (CS) and an Internal Hex connection (IH). the fixture has a straight coronal part, a slightly tapered body and a conical apical part. We will use MultiNeO CS in control group. One of the MultiNeO biggest clinical advantages since it is as good at bone type 4 as it is at bone type 1, 2 or 3.

Topography and surface roughness of MultiNeO lead to some clinical advantages:

Increased early BIC; Increased primary and secondary stability; Shortened healing period; Accelerated and improved osseointegration process.

MultiNeO CS has an implant surface similar to the aforementioned SLA surface manufactured by Straumann. In fact, SLA is a sub-micron scale roughness created by Aluminum oxide blasting and double acid etching.

NINA- MultiNeO NH is used for treatment group, and it is being tested. NINA MultiNeO NH has got an innovative bioactive surface.

NINA MultiNeO NH surface is a combination of the abovementioned roughening process and the creation of titanium oxide nano structure. Its hydrophilic part is created by resorbable salt thus maintaining its hydrophilicity.

Although a variety of implant surface are available for implant rehabilitation, the first hypothesis is that NINA MultiNeO NH Alpha-Bio Tec ® will be positively adopted for rehabilitation of missing teeth with shorter healing time and less marginal bone loss.

The idea behind these studies is to maximize the effect of the bioactive surface testing its behavior in a poor host environment with a reduced time

ELIGIBILITY:
Inclusion Criteria:

1. Patient with type 1-2 post extraction sites
2. Subject is 30-80 years old
3. Patient ASA 1 or 2
4. Patients with healthy periodontal conditions (Treated periodontitis, PI<25%, BoP<25%)
5. Patients that are willing to sign an informed consent and participate in a clinical study

Exclusion Criteria:

1. Absence Type 1-2 post extraction sites
2. Patient ASA 3 or 4
3. Untreated Periodontitis
4. Any sites where an implant already failed sites
5. Allergy declared to one or more medicaments to be used during treatment
6. Pregnancy (confirmed by verbal inquiry)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | 6 months after implant placement
  Radiographic evaluation of the marignal bone level around the implant using a periapical x ray. marginal bone loss is in millimeters and indicates how many millimeters of bone has been lost
Marginal bone loss | 12 months after implant placement
  Radiographic evaluation of the marignal bone level around the implant using a periapical x ray. marginal bone loss is in millimeters and indicates how many millimeters of bone has been lost
Implant stability | immediately after implant placement
  check implant stability using resonant frequency analysis (RFA)
Implant stability | 30 days after implant placement
  check implant stability using resonant frequency analysis (RFA)
Implant stability | 45 days after implant placement
  check implant stability using resonant frequency analysis (RFA)

SECONDARY OUTCOMES:
insertion torque curve | During implant placement (T0 baseline)
  The Insertion torque data were recorded and exported as a curve The torque curve records the amount of energy that was needed for arrive at the positioning of the implant.
  unit of measurement of torque is Newton centimeter (Ncm)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Canullo, DDS PhD, Principal Investigator — Studio odontoiatrico associato Cicchese Canullo
Locations (1):
- Studio Odont.Associato Dr.P.Cicchese E L.Canullo, Rome, Italy/Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Clinical data will be first recorded in EDC (electronic data capture). Then data will be entered into one-central computerized database.
  Patient adverse events will be reported, including during implant placement and throughout follow-up period.
  Implant details parameters and data will be recorded into EDC. The data then will be entered into one central computerized database and analyzed statistically for evaluation of the results.
  The study database will be designed and maintained using Microsoft Excel. an identification code will be assigned to each patient
Supporting Information: Study Protocol, SAP, CSR
Time Frame: the data will be available for the duration of the study
Access Criteria: the data will be available for the duration of the study

REFERENCES:
- [Background] Wennerberg A, Albrektsson T. Effects of titanium surface topography on bone integration: a systematic review. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:172-84. doi: 10.1111/j.1600-0501.2009.01775.x. PMID 19663964
- [Background] Han J, Lulic M, Lang NP. Factors influencing resonance frequency analysis assessed by Osstell mentor during implant tissue integration: II. Implant surface modifications and implant diameter. Clin Oral Implants Res. 2010 Jun;21(6):605-11. doi: 10.1111/j.1600-0501.2009.01909.x. PMID 20666787
- [Background] Gianfreda F, Antonacci D, Raffone C, Muzzi M, Pistilli V, Bollero P. Microscopic Characterization of Bioactivate Implant Surfaces: Increasing Wettability Using Salts and Dry Technology. Materials (Basel). 2021 May 17;14(10):2608. doi: 10.3390/ma14102608. PMID 34067747